CLINICAL TRIAL: NCT04437134
Title: On-line Neuromuscular Exercise and Education for Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Slagelse Hospital (Other)
Collaborators: Region Zealand (Other)
Responsible Party: Principal Investigator, Pætur Mikal Holm, Physiotherapist, PhD, Postdoc., Slagelse Hospital
Other Study IDs: SlagelseH; J.nr. 20-000013 (Other: Scientific Ethics Committee of Region Zealand)
Record Dates: First submitted 2020-06-07; First posted 2020-06-18 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Exercise; Education; On-line; Pain; Function; Quality of Life
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity; Pain | interventions — Educational Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- On-line exercise and education: Exercise (12 sessions) and education (2-3 sessions) delivered on-line. Patients attend both the exercise and educational sessions by logging on to virtual rooms using links sent out by e-mail. The sessions are led and supervised by GLA:D certified physiotherapists.
  Interventions: Other: On-line exercise and education
- On-site exercise and education: Exercise (12 sessions) and education (2-3 sessions) delivered on-site. Patients attend both the exercise and educational sessions at physiotherapy clinics in Denmark. The sessions are led and supervised by GLA:D certified physiotherapists.
  Interventions: Other: On-site exercise and education

INTERVENTIONS:
Other: On-line exercise and education — Exercise:
  Exercise is performed twice weekly for 6 weeks. Each exercise session lasts approximately 60 min. and consists of three parts; warm-up (10 min.), neuromuscular exercises (40 min.), and cool-down/stretching (10 min.). The neuromuscular exercises include exercises for core stability, postural orientation, function and leg muscle strength. Exercises are performed in 2-3 sets with 10-15 repetitions with three levels of difficulty described. The exercises follow the standardized GLA:D exercise protocol. Patients are instructed in how to use alternative equipment at home for each exercise if necessary prior to the first on-line exercise session.
  Education:
  Patients attend two to three on-line educational sessions at the start of each GLA:D program. The educational sessions focus on disease-management and self-help strategies, including OA disease features and symptoms, treatment options, and exercise and physical activity as treatment.
  Groups: On-line exercise and education
Other: On-site exercise and education — Exercise:
  Exercise is performed twice weekly for 6 weeks. Each exercise session lasts approximately 60 min. and consists of three parts; warm-up (10 min.), neuromuscular exercises (40 min.), and cool-down/stretching (10 min.). The neuromuscular exercises include exercises for core stability, postural orientation, function and leg muscle strength. Exercises are performed in 2-3 sets with 10-15 repetitions with three levels of difficulty described. The exercises follow the standardized GLA:D exercise protocol. The exercise sessions are delivered at physiotherapy clinics in Denmark.
  Education:
  Patients attend two to three on-site educational sessions at the start of each GLA:D program. The educational sessions focus on disease-management and self-help strategies, The educational sessions focus on disease-management and self-help strategies, including OA disease features and symptoms, treatment options, and exercise and physical activity as treatment.
  Groups: On-site exercise and education

SUMMARY:
Due to enforced social distancing as a direct consequence of the COVID-19 pandemic, many on-site health care services are unavailable. This study seeks to investigate the relative effectiveness of an alternative on-line delivery model of exercise and education compared to on-site delivery in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Due to the extraordinary events of the 2020 COVID-19 pandemic, finding alternative delivery-models of treatment has come to the forefront of public health services worldwide. Consequently, on-line treatment is rapidly becoming an integral part of public health service. For patients with knee osteoarthritis (OA), where non-pharmacological and non-surgical treatment is considered first-line treatment, on-line delivered exercise has already shown promise and may be a viable treatment option, especially when traditional on-site exercise delivery models are unavailable. However, further studies are needed to clarify the relative effectiveness of on-line exercise and education when compared to on-site exercise and education programs.

This study aims to evaluate the effects of on-line exercise and education in knee OA compared to a cohort of similar knee OA patients completing the same exercise and education program through on-site delivery.

This study includes two cohorts of knee OA patients receiving the same exercise and education program through different delivery models (on-line vs. on-site). The on-line cohort is a new treatment delivery initiative, born out of the COVID-19 enforced shutdown of all non-critical on-site health care. The on-site cohort is comprised of knee OA patients from a patient registry, collecting outcome data as part of the exercise and education program.

The exercise and education program is called Good Life with osteoArthritis in Denmark (GLA:D), and consists of two to three disease-specific educational sessions and 12 neuromuscular exercise sessions (NEMEX-TJR). GLA:D originates from Denmark and has currently been implemented in Australia, Canada, China, Switzerland and New Zealand.

This study will primarily compare outcomes of pain, function and quality of life between the two different treatment delivery models and will provide important insights in effectiveness of alternative delivery models of recommended first-line care for patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Knee OA symptoms resulting in contact with the health care system

Exclusion criteria (both study groups):

* Another reason than OA for the problems; includes tumour or inflammatory joint disease
* Other symptoms that are more pronounced than the OA symptoms; i.e. chronic, generalised pain or fibromyalgia.

In addition, for the on-line study group:

* Previous participation in similar exercise and education programs (i.e. the on-site version)
* Lack of necessary equipment or skills to administer on-line participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included into this study are adults, reporting knee OA symptoms as their main source of pain.
  Both study groups (on-line and on-site exercise and education) are comprised of patients with symptomatically verified (all) and radiographically verified (most) knee OA.
  On-line exercise and education:
  Patients referred for assessment in secondary care due to knee OA symptoms.
  On-site exercise and education:
  Patients with knee OA symptoms referred to a physiotherapist either by their general practitioner, by an orthopedic surgeon, or by self-referral.
Sampling Method: Non-Probability Sample
Enrollment: 3789 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Knee impact summary | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Summary score from the Knee injury and Osteoarthritis Outcome Score, short version (KOOS 12). The summary score is calculated as the average score from the KOOS 12 subscales pain, function and quality of life (QOL), ranging from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Fast-paced walking ability | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months)
  Fast-paced walking ability is recorded by the physiotherapists and evaluated using the 40-m fast-paced walk test.
Chair-stand ability | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months)
  Chair-stand ability is recorded by the physiotherapists and evaluated using the 30-s chair-stand test.
Self-reported function | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report of function during daily life using the subscale function from the KOOS 12 questionnaire with scores ranging from 0 (worst) to 100 (best).
Self-reported pain | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report of pain using the subscale pain from the KOOS 12 questionnaire with scores ranging from 0 (worst) to 100 (best).
Self-reported quality of life | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report of quality of life using the subscale quality of life from the KOOS 12 questionnaire with scores ranging from 0 (worst) to 100 (best).
Pain intensity | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Mean pain intensity during the last week in the most affected knee is evaluated on a 100 mm visual analogue scale (VAS) with terminal descriptors of 'no pain' (0 mm) and 'maximum pain' (100 mm).
Physical activity and exercise | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report of time spent (frequency and duration) on structured physical activity and exercise.

OTHER OUTCOMES:
Patient satisfaction | Primary follow-up point: Completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report of satisfaction with the GLA:D program.
Continuation of exercise | Follow-up point: 12 months
  Patients self-reporting if, how and where they have continued exercising.
Self-reported activity levels | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report their current activity levels using the University of California, Los Angeles (UCLA) activity scale, ranging from 1 (inactive, dependent on others) to 10 (regular participation in high-impact sports).
Usage of what was learned during GLA:D | Primary follow-up point: Completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report of use of acquired skills and knowledge from the GLA:D program.
Symptom management | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report of how they handle flare-ups in their knee OA symptoms.
Intake of pain killers | Primary follow-up: Change from baseline to completion of GLA:D program (an average of three months).
  Intake of painkillers is evaluated by the physiotherapist asking the patients about intake of any joint related medication. If taking painkillers, the patients are asked which type and whether or not they were taken because of their knee pain.
Sick leave | Follow-up points: Baseline and 12 months
  Patients self-report of sick leave due to knee symptoms.
Health-related quality of life, index score | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report of their health situation using EuroQol, 5 dimensions, 5 levels (EQ-5D-5L) score (-0.624 to 1; worst to best).
Health-related quality of life, visual analogue scale | Primary follow-up point: Change from baseline to completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report of their health situation using the EuroQol visual analogue scale (EQ VAS), ranging from 0-100 (worst to best).
Global perceived effect | Primary follow-up point: Completion of GLA:D program (an average of three months). Secondary follow-up point: 12 months
  Patients self-report of current knee condition compared to before participation in GLA:D, scored on a 7-point likert scale (much worse to much better).
Pain during exercise (only for on-line group) | Immediately prior to, and immediately after each exercise session
  Patients self-report of pain during each exercise session, rated using a numeric pain rating scale (NPRS) 0-10, with zero representing no pain and 10 representing extreme pain.

CONTACTS AND LOCATIONS:
Overall Officials: Pætur M Holm, PhD, Principal Investigator — Department of Physiotherapy and Occupational Therapy; Søren T Skou, Professor, Study Chair — Department of Physiotherapy and occupational Therapy
Locations (4):
- Denmark (4):
  - Department of Orthopedic Surgery, Næstved-Slagelse-Ringsted Hospitals, Næstved, Region Sjælland
  - Department of Physiotherapy and Occupational Therapy, Næstved-Slagelse-Ringsted Hospitals, Næstved, Region Sjælland
  - Department of Physiotherapy and Occupational Therapy, Næstved-Slagelse-Ringsted Hospitals, Slagelse, Region Sjælland
  - University of Southern Denmark, Odense, Region Southern Denmark

IPD SHARING:
Plan to Share IPD: Undecided